CLINICAL TRIAL: NCT01323764
Title: A Double- Blinded Comparison of the Accuracy of ShuntCheck, a Non-Invasive Device, to Radionuclide Shunt Patency Test in Evaluating Shunt Function in Patients With Adult Hydrocephalus With Possible Shunt Obstruction
Brief Title: ShuntCheck Versus Radionuclide in Evaluating Shunt Function in Symptomatic NPH Patients
Acronym: SCNPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NeuroDx Development (Industry)
Collaborators: Sinai Hospital of Baltimore (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NDxDev-SCMP-2012; R43NS067770-01A1 (NIH)
Record Dates: First submitted 2011-03-21; First posted 2011-03-28 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; CSF shunts; Normal Pressure Hydrocephalus; NPH; ShuntCheck; Shunt Malfunction; Suspected shunt malfunction in adult hydrocephalus patients
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radionuclide SPS (Active Comparator): Radionuclide Shunt Patency Study
  Interventions: Device: ShuntCheck test

INTERVENTIONS:
Device: ShuntCheck test — Non-invasive, thermal dilution test for CSF shunt flow compared to radionuclide shunt patency testing
  Other Names: ShuntCheck

SUMMARY:
The purpose of this study is to compare the accuracy of ShuntCheck (SC) and ShuntCheck plus Micro-Pumper (SC+MP) to radionuclide shunt patency testing (SPS) in evaluating shunt function in patients with adult hydrocephalus (AH) implanted with ventriculoperitoneal (VP) shunts when shunt obstruction is suspected and a diagnostic procedure such as radionuclide shunt patency testing (SPS) is required.

DETAILED DESCRIPTION:
The primary objective is to demonstrate that the accuracy of SC and SC+MP for determining whether a VP shunt is patent or obstructed is statistically no different than the accuracy of the accepted standard test, radionuclide shunt patency study, when performed simultaneously.

A secondary objective is to determine SC and SC+MP results in the presence of possible partial obstruction, which defined as subjects with radionuclide clearance measured by T1/2 of 8 to 10 minutes.

A secondary objective is to compare ShuntCheck flow rate results to simultaneous radionuclide clearance as measured by T1/2. A secondary objective is to demonstrate that ShuntCheck flow rate results are statistically equivalent to simultaneous radionuclide clearance measured by T1/2

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women > 35 years of age;
2. Capable of providing valid signed informed consent, or has a legal guardian, health care agent, or surrogate decision maker (according to local statutes, and collectively referred to as "surrogates" in this protocol) capable of providing valid, signed informed consent;
3. Possess a shunt placed for AH;
4. A radionuclide shunt patency study has been ordered because of suspected shunt obstruction
5. Subject is willing and able to return to the treating physician for evaluation of the outcome of the shunt patency study

Exclusion Criteria:

1. Presence of multiple shunts, or presence of more than one distal shunt catheter (regardless of function) crossing the clavicle ipsilateral to the shunt with suspected obstruction;
2. ShuntCheck test would interfere with standard patient care, or emergency shunt surgery that cannot be delayed is indicated;
3. Presence of an interfering open wound or edema over any portion of the VP shunt;
4. Subject is unwilling or unable to return to the treating physician for the SPS and ShuntCheck testing.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of ShuntCheck vs SPS | Day 1
  The primary efficacy objective is the sensitivity and specificity of the ShuntCheck test.
  The performance of ShuntCheck test will be compared to the radionuclide scanning done on the day of ShuntCheck administration. Primary efficacy of the SC and SC+MP test will be determined by comparing SC and SC+MP performance to results of radionuclide scanning according to a standard 2 x 2 table, with a Positive test result defined as evidence of shunt obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Williams, MD, Principal Investigator — Sinai Hospital of Baltimore, LifeBridge Health; Sherman C Stein, MD, Study Chair — NeuroDx Development; Marek Swoboda, PhD, Study Director — NeuroDx Development
Locations (1):
- Sinai Hospital of Baltimore, LifeBridge Health, Baltimore, Maryland, United States